CLINICAL TRIAL: NCT06566274
Title: Clinical Efficacy and Safety Evaluation of Thumbtack Needle in Nausea and Vomiting in Pregnancy: a Randomized Controlled Clinical Trial
Brief Title: Thumbtack Needle in the Treatment of NVP
Acronym: TN-NVP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dongmei Huang (Other)
Responsible Party: Sponsor-Investigator, Dongmei Huang, associate professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN-NVP
Record Dates: First submitted 2024-08-12; First posted 2024-08-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Nausea and Vomiting in Pregnancy (NVP)
Keywords: Nausea and vomiting in pregnancy; Thumbtack needle
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thumbtack needle (TN) group (Active Comparator): The main acupoints of treatment are Zhongwan (CV12), bilateral Neiguan (SP6), and bilateral Zusanli (ST36), with a total of 5 acupoints. patients with Qi stagnation should be added Danzhong (CV17) or Ashi acupoint (the most prominent tender point between CV 17 and CV12), patients with liver and stomach disharmony should be added bilateral BL17, patients with phlegm-dampness obstruction should be added bilateral ST40, and patients with weak spleen and stomach should be added bilateral BL21. The above acupoints are treated with TN. The TN will be reserved in the acupoints for 3 days. During the 3-day retention of TN, the patient presses the TN 3 times a day and half a minute per time per acupoint. After 3 days of retention of TN, the patient is instructed to go to the hospital and receive the next TN treatment. A total of 5 treatments were applied for a duration of 15 days.
  Interventions: Device: thumbtack needle
- sham TN group (Sham Comparator): The acupoints of sham TN group are the same as those of TN group. The use of sham TN was the same as that of the TN group. During the 3-day retention of sham TN, the patients are asked not to press them. After 3 days retention of sham TN, the patient was instructed to go to the hospital, where the doctor removed the sham TN, and conducted the next treatment after local skin disinfection. A total of 5 treatments were given for a duration of 15 days.
  Interventions: Device: sham thumbtack needle

INTERVENTIONS:
Device: thumbtack needle — As a kind of intradermal needle, thumbtack needle (TN) is a method of shallow puncture and long-term needle.After the TN is attached into the acupoints, it will be reserved in the acupoints for 3 days. After 3 days of retention of TN, the patient is instructed to go to the hospital, where the doctor removes the needle, disinfect the local skin of acupoints and conducts the next TN treatment. A total of 5 treatments were applied for a duration of 15 days.
  Arms: thumbtack needle (TN) group
Device: sham thumbtack needle — The sham TN used in the sham TN group has no needle body and its appearance and shape are similar to the real TN. But it does not produce a needle-like effect.
  The acupoints of sham TN group are the same as those of TN group. The use of sham TN is the same as that of the TN group. After 3 days retention of sham TN, the patient will be instructed to go to the hospital, where the doctor remove the sham TN, and conduct the next treatment after local skin disinfection. A total of 5 treatments will be applied for a duration of 15 days.
  Arms: sham TN group

SUMMARY:
This project intends to use multi-center, large-sample, randomized, controlled, blinded clinical trials to observe the clinical efficacy and safety of thumbtack needle (TN) on nausea and vomiting in pregnancy (NVP).

DETAILED DESCRIPTION:
Nausea and vomiting in pregnancy (NVP) is the most common and intractable problem in the first trimester and is the second most common presentation during pregnancy. All types of NVP affect the quality of life of pregnant women, and the intensity of influence increases with the frequency of symptoms. Due to the lack of awareness of NVP and the concern about the teratogenicity of drugs to embryos, the treatment of NVP is always insufficient, and the choice of drug regimen is conservative.

Acupuncture using traditional millineedle is effective on NVP, however, it is generally painful when the millineedle is inserted into the body, and the needling sensation of soreness, numbness, swelling and pain during acupuncture is sometimes beyond patient's acceptability, or even produce adverse effects on pregnancy. Moreover, patients may have to visit acupuncturist daily using millineedle, which may causes high financial costs and reduce the medial adherence. Therefore, although acupuncture with millineedle is effective on NVP, its application in clinical practice is still very limited.

As a kind of intradermal needle, thumbtack needle (TN) is a method of shallow puncture and long-term retention needle. Although the amount of stimulation of TN is weaker than that of millineedle, it has a much longer effect and can produce continuous and stable stimulation, and therefore, its cumulative effect is often better than that of traditional millineedle acupuncture. Moreover, due to the tiny needle body of TN (the diameter of the needle body is only 0.15 ~ 0.25mm, and the length of the needle body is only 1.2 ~ 2.5mm), it will not hurt the subcutaneous nerves, blood vessels, viscera and other tissues, which is very comfortable and safe to treat, and overcomes the needle sting pain of traditional millineedles. However, up to now, it is unknown whether TN can produce the same effect as the acupuncture in NVP.

This project is a multi-center, large-sample and blinded RCT designed to collect the highest quality evidence of complete data, including nausea and vomiting, quality of life, anxiety and depression, weight change, blood electrolyte levels, liver and kidney function, thyroid function, intravenous fluid treatment, use of additional drugs, hospital admission, pregnancy complications (gestational diabetes and hypertensive diseases), pregnancy outcomes and neonatal outcomes in women with VNP.

ELIGIBILITY:
Inclusion Criteria:

* The mother's age is 20 ~ 45 years old, the gestational age is 6 ~ 12 weeks, and the ultrasound confirms that it is an intrauterine single or multiple pregnancy, and the weight loss is less than 10% compared with before pregnancy.
* Women diagnosed with moderate to severe NVP in the first trimester: the severity of NVP was determined by the PUQE score (see Table 1), and the PUQE score ranged from 3 ~ 15, < 6 was mild NVP, 6 ~ 12 was moderate NVP, and ≥13 was severe NVP. PUQE score ≥ 6 may be included in this study.
* Women voluntarily sign the informed consent form.

Exclusion Criteria:

* Age >20 years, and <45 years.
* Gestational > 6 weeks, or <12 weeks.
* PUQE score <6.
* frequent nausea and vomiting, weight loss of >10% compared with before pregnancy; or symptoms such as listlessness, paleness, dry skin, sunken eye sockets, and a marked decrease in urine output (less than 400ml of urine in 24 hours or less than 5 times and a small amount of urine in 24 hours).
* At rest, body temperature > 38°C, systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 60 mmHg or > 90 mmHg, heart rate ≥ 100 beats per minute, or oxygen saturation < 95%.
* Urinalysis: urine ketones: +++ and above; or (and) urine protein: ++ and above.
* Blood biochemistry: serum potassium≤3.0mmol/L, serum sodium≤130mmol/L; or abnormal liver function: elevated liver enzymes ≥ 2 times the upper limit of normal; or renal dysfunction: elevated serum creatinine and urea nitrogen.
* Other digestive diseases that cause nausea and vomiting, such as gastrointestinal infections (with diarrhea), gastric ulcers (with epigastric pain or hematemesis), cholecystitis, biliary roundworms, pancreatitis (with abdominal pain, plasma amylase levels rise to 5 ~ 10 times normal), viral hepatitis (positive hepatitis virology, liver enzyme levels ≥ 1 000 U/L) or acute fatty liver during pregnancy, tumors of the digestive tract.
* Suffering from immune diseases such as systemic lupus erythematosus, scleroderma, dermatomyositis, IgG4-related diseases, immune nephropathy, etc.
* Have uncorrected diseases of the endocrine system, such as diabetes, Addison's disease, hyperthyroidism, hypothyroidism, thyroid tumors, adrenal tumors, etc.
* Suffering from neurological diseases such as migraine, neuromyelitis optica, epilepsy, neurologic tumors, etc.
* In the past 1 week, have taken antiemetic drugs such as ondansetron, metoclopramide (metoclopramide), promethazine, anti-vomiting Chinese medicine, etc.
* Monoamine oxidase inhibitors are used.
* Have received TN treatment in recent 3 months.
* Unwilling to sign the informed consent of this study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Score change of pregnancy unique quantification of emesis (PUQE) scale from baseline to day 15. | Baseline to day 15
  PUQE scores ranged 3 to 15, with higher scores indicating a worse outcome. PUQE scores were evaluated before treatment and on days 3, 6, 9, 12, and 15 of treatment. The primary outcome measure was the change of PUQE score from baseline to day 15.

SECONDARY OUTCOMES:
The Nausea and Vomiting of Pregnancy Quality of Life (NVPQOL) questionnaire | Baseline to day 15
  The NVPQOL range 30-210, with higher scores means a worse quality of life
Anxiety status survey: Zung-SAS | Baseline to day 15
  Zung-SAS range 25-100, with higher scores means more severe anxiety
Depression status survey: Zung-SDS | Baseline to day 15
  Zung-SDS range 20-80, with higher scores means more severe depression
Sleep status survey: The Pittsburgh sleep quality index (PSQI) | Baseline to day 15
  PSQI range 0-21, with higher scores means poorer sleep status
Change of maternal weight from baseline to last visit | Baseline to day 15
  Change of maternal weight from baseline to the last visit
Change of electrolyte index (sodium) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of electrolyte index (potassium) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of electrolyte index (calcium) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of electrolyte index (chlorine) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of electrolyte index (phosphorus) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of electrolyte index (magnesium) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of electrolyte index (iron) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: μmol/L
Change of electrolyte index (zinc) | Baseline to day 15
  Value changes from baseline to the last visit. Unit: μmol/L
Carbon dioxide combining power in the blood | Baseline to day 15
  carbon dioxide conbining power in the artery blood. Unit: mmol/L
Change of AST | Baseline to day 15
  Value changes from baseline to the last visit. Unit: U/L
Change of ALT | Baseline to day 15
  Value changes from baseline to the last visit. Unit: U/L
Change of ALP | Baseline to day 15
  Value changes from baseline to the last visit. Unit: U/L
Change of creatinine | Baseline to day 15
  Value changes from baseline to the last visit. Unit: μmol/L
Change of urea | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mmol/L
Change of TSH | Baseline to day 15
  Value changes from baseline to the last visit. Unit: mIU/L
Change of free triiodothyronine | Baseline to day 15
  Value changes from baseline to last visit. Unit: pmol/L
Change of free thyroxine | Baseline to day 15
  Value changes from baseline to the last visit. Unit: pmol/L
Change of cortisol | Baseline to day 15
  Value changes from baseline to the last visit. Unit: ug/dL
Change of ghrelin | Baseline to day 15
  Value changes from baseline to the last visit. Unit: ng/ml
Change of leptin | Baseline to day 15
  Value changes from baseline to the last visit. Unit: ng/ml
Change of 5-hydroxytryptamine | Baseline to day 15
  Value changes from baseline to the last visit. Unit: ng/ml
Change of substance P | Baseline to day 15
  Value changes from baseline to the last visit. Unit: pg/ml
Change of arginine vasopressin plasma | Baseline to day 15
  Value changes from baseline to the last visit. Unit: pg/ml
Change of GDF 15 | Baseline to day 15
  Value changes from baseline to the last visit. Unit: pg/ml
Change of IGFBP 7 | Baseline to day 15
  Value changes from baseline to the last visit. Unit: ng/ml
Number of participants with intravenous fluid treatment during treatment | Baseline to day 15
  If the patient suffers from dehydration or electrolyte imbalances, intravenous fluid treatment will be done.
Number of participants with concomitant treatment | Baseline to day 15
  How many participants with concomitant treatment
Number of participants with hospital admission during treatment | Baseline to day 15
  If the patient suffers from further aggravation of neasua and vomiting or hyperemesis gravidarum, hospital admission will be done.
Number of participants with termination of pregnancy | Data collected from baseline to 1 week after termination of pregnancy
  If the patient suffers from further aggravation of hyperemesis gravidarum, the termination of a wanted pregnancy will be done due to life in danger. Or if congenital anomalies are found by ultrasound, the termination of a wanted pregnancy will be done.
Pregnancy complications | Data collected from baseline up to 42 days after parturition
  Pregnancy complications including miscarriage (in the first trimester and in the second trimester), hypertensive disorders, gestational diabetes and so on.
Number of participants with preterm birth | Data collected from baseline to 42 days after postpartum
  How many participants with preterm birth
Delivery outcomes | Data collected from baseline to 42 days after postpartum
  Delivery outcomes including live birth, vaginal birth, caesarean section, gestational age, etc.
Number of participants with neonatal congenital anomalies | Data collected from baseline to 42 days after postpartum.
  Participants with neonatal congenital anomalies
Number of participants with neonatal mortality | Data collected from baseline to 42 days after postpartum.
  Participants with neonatal mortality
Number of participants with neonatal hypoglycemia | From baseline to 42 days after postpartum.
  Participants with neonatal hypoglycemia.
Number of participants with neonatal NICU admission. | From baseline to 42 days after postpartum.
  Participants with neonatal NICU admission.
Patient's satisfaction with treatment | Baseline to day 15
  Questionnaire such as loss of confidence, doubt of the efficacy or intolerance to the treatment of TTN and so on. The answer is "yes" or "no".
Patient's compliance with treatment | Baseline to 42 days after postpartum.
  The percentage of the participants which finish the treatment and the follow-up.
Adverse events and serious adverse events | Baseline to the end of follow-up (four weeks after the end of treatment)
  The percentage of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Huang, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (13):
- China (13):
  - Jingzhou Hospital of Traditional Chinese Medicine, Jingzhou, Hubei
  - Nanzhang County Traditional Chinese Medicine Hospital, Nanzhang Chengguanzhen, Hubei
  - Qianjiang Central Hospital, Qianjiang, Hubei
  - Qianjiang Maternal and Child Health Care Hospital, Qianjiang, Hubei
  - Shiyan People's Hospital, Shiyan, Hubei
  - Suizhou Maternal and Child Health Care Hospital, Suizhou, Hubei
  - Wuhan Jinxin Gynecology and Obstetrics Hospital of Integrative Medicine, Wuhan, Hubei
  - Department of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Hospital of Traditional Chinese Medicine, Xiangyang, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiaogan Maternal and Child Health Care Hospital, Xiaogan, Hubei
  - Dongchangfu District Maternal and Child Health Care Hospital of Liaocheng City, Liaocheng, Shandong
  - Aksu Prefecture Maternal and Child Health Hospital, Aksu, Xinjiang

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-09-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT06566274/Prot_000.pdf
  • Informed Consent Form (2024-09-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT06566274/ICF_001.pdf